CLINICAL TRIAL: NCT03061474
Title: A Double-Blind-Randomized, Placebo-Controlled Adaptive Design Trial of Nicotinamide in Mild Cognitive Impairment Due to Alzheimer's Disease and Mild Alzheimer's Disease Dementia
Brief Title: Nicotinamide as an Early Alzheimer's Disease Treatment
Acronym: NEAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Joshua Grill, Associate Professor, Psychiatry & Human Behavior, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20163246
Record Dates: First submitted 2017-02-13; First posted 2017-02-23 (Actual); Results first posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-09

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Alzheimer's Disease; Nicotinamide; Niacinamide; Niacin; Nicotinic Acids; Vitamin; Neurodegenerative Diseases; Tauopathies; Dementia
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Neurodegenerative Diseases; Tauopathies; Dementia | interventions — Niacinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blind-Randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nicotinamide (Experimental): 1500mg twice daily: 2, 750mg tablets taken orally twice daily
  Interventions: Drug: Nicotinamide
- Placebo (Placebo Comparator): 1500mg twice daily: 2, 750mg tablets taken orally twice daily
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Nicotinamide — Niacinamide (nicotinamide; 99%) is produced in a 750 mg sustained release tablet.
  Other Names: Niacinamide
  Arms: Nicotinamide
Drug: Placebo Comparator — Oral Tablet
  Arms: Placebo

SUMMARY:
The purpose of this research study is to test whether nicotinamide, also known as vitamin B3 or niacinamide, taken in high doses, can reduce phosphorylation of tau (the protein that accumulates in neurofibrillary tangles) in people with Mild Cognitive Impairment or mild Alzheimer's disease (AD) dementia.

DETAILED DESCRIPTION:
Nicotinamide, the amide of nicotinic acid (vitamin B3/niacin), is an oral therapy with a wealth of clinical data in a variety of therapeutic areas, including preliminary data supporting its safety in Alzheimer's disease (AD). Preclinical work in a mouse model that develops both plaques and tangles supports the hypothesis that nicotinamide can act as a histone deacetylase (HDAC) inhibitor to reduce phosphorylation of tau.

The study will implement a group sequential design, incorporating a futility analysis with a go/no-go decision conditional on cerebral spinal fluid CSF biomarker outcomes at 12-months. The primary outcome for the trial is change in p-tau231.

This study timeline includes a screening phase of up to 60 days and treatment phase which is expected to last about 48 weeks and will include 4 study visits.

An additional 12-month treatment and follow-up period is planned, contingent upon a "go" decision based on the primary outcome (CSF p-tau231) or one planned secondary outcome (CSF p-tau181)

ELIGIBILITY:
Inclusion Criteria:

1. Mild Cognitive Impairment (MCI) or dementia due to Alzheimer's disease (AD)
2. Biomarker criteria:

   Cerebral Spinal Fluid (CSF) Amyloid Beta 1-42 (Aβ42) <= 600 pg/mL, or A ratio of total tau to Aβ42 ≥ 0.39.
3. Mini-Mental State Exam (MMSE) ≥ 20
4. Blood laboratories, urinalysis, and electrocardiogram are within normal limits or deemed clinically not significant by the site investigator
5. Stable medications (including approved AD therapies) for at least 4 weeks
6. At least 6 years of education
7. Able to swallow oral tablets
8. Speaks English fluently
9. Available qualified study partner (≥3 times per week in-person communication with the participant)

Exclusion Criteria:

1. Active neurological or psychiatric diagnosis other than AD that may affect cognition and/or function. (Obstructive sleep apnea is permitted, if treated.)
2. Inability to undergo lumbar puncture, including use of Coumadin, novel oral anticoagulants, clopidogrel, or dipyridamole. Use of aspirin <= 325mg daily is permitted.
3. Hachinski ischemic scale > 4
4. Magnetic Resonance Imaging (MRI) incompatibility
5. MRI evidence of cortical stroke >1cm, superficial siderosis, or extensive white matter hyperintensity (Cardiovascular Health Study score 7-8+)
6. Diagnosis of cancer in the previous 5 years (with the exception of basal or squamous cell carcinoma)
7. Geriatric Depression Scale (GDS) score >6
8. History within the past 5 years of alcohol or substance use disorder
9. Laboratory evidence of a clinically significant abnormality that may interfere with study assessments
10. Active partial or total malabsorptive disease (e.g., celiac disease)
11. Resides in a skilled nursing facility
12. Participation in a clinical trial of a potential disease-modifying therapy for AD in previous 6-months (time between last investigational drug administration and baseline for the current study)
13. Pregnant, lactating or of child bearing potential (that is, women must be 2 years post-menopausal or surgically sterile to be considered not child bearing potential).
14. Unwillingness to abstain from over-the-counter nicotinamide for the duration of the trial

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Grill, Ph.D., Principal Investigator — Associate Professor of Psychiatry and Human Behavior
Locations (2):
- United States (2):
  - University of California, Irvine, Irvine, California
  - University of California, Los Angeles, Los Angeles, California

IPD SHARING:
Plan to Share IPD: Yes
Data sharing is integral to the ADCS's mission to develop and execute innovative clinical trials focused on interventions that may prevent, delay, or treat the expression of Alzheimer's disease and related dementias. The ADCS is committed to sharing resources and tools, including data, biospecimens, trial designs, outcome and analysis measures following NIH guidelines.
  DATA Sharing: The ADCS Data and Sample Sharing Committee (DSSC) grants access to de-identified data to individuals who complete the request process and agree to the conditions in an ADCS/UCSD Data Us Agreement (DUA). After approval and receipt of the fully executed DUA, applicants are authorized to acquire data. Non-compliance with the DUA, including the requirement to provide requested updates will jeopardize further access to data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after publication
Access Criteria: Data requestors must complete ADCS data and sample sharing request form. Upon approval, requestors must complete a data use agreement prior to accessing data.
URL: https://www.adcs.org/data-sharing

REFERENCES:
- [Background] Green KN, Steffan JS, Martinez-Coria H, Sun X, Schreiber SS, Thompson LM, LaFerla FM. Nicotinamide restores cognition in Alzheimer's disease transgenic mice via a mechanism involving sirtuin inhibition and selective reduction of Thr231-phosphotau. J Neurosci. 2008 Nov 5;28(45):11500-10. doi: 10.1523/JNEUROSCI.3203-08.2008. PMID 18987186
- [Background] Liu D, Pitta M, Jiang H, Lee JH, Zhang G, Chen X, Kawamoto EM, Mattson MP. Nicotinamide forestalls pathology and cognitive decline in Alzheimer mice: evidence for improved neuronal bioenergetics and autophagy procession. Neurobiol Aging. 2013 Jun;34(6):1564-80. doi: 10.1016/j.neurobiolaging.2012.11.020. Epub 2012 Dec 25. PMID 23273573
- [Derived] Ketron GL, Grun F, Grill JD, Feldman HH, Rissman RA, Brewer GJ. Pharmacokinetic and pharmacodynamic assessment of oral nicotinamide in the NEAT clinical trial for early Alzheimer's disease. Alzheimers Res Ther. 2025 Mar 11;17(1):59. doi: 10.1186/s13195-025-01693-y. PMID 40069789
- [Derived] Grill JD, Tam S, Thai G, Vides B, Pierce AL, Green K, Gillen DL, Teng E, Kremen S, Beigi M, Rissman RA, Leger GC, Balasubramanian A, Revta C, Morrison R, Jennings R, Pa J, Zhang J, Jin S, Messer K, Feldman HH. Phase 2A Proof-of-Concept Double-Blind, Randomized, Placebo-Controlled Trial of Nicotinamide in Early Alzheimer Disease. Neurology. 2025 Jan 14;104(1):e210152. doi: 10.1212/WNL.0000000000210152. Epub 2024 Dec 13. PMID 39671543

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 46 participants received at least 1 dose of study drug.
Period: Overall Study
Arm/Group | Nicotinamide | Placebo
Started | 24 | 22 (22 participants received treatment therapy.)
Completed | 22 | 18
Not Completed | 2 | 4
Not completed — Adverse Event | 2 | 0
Not completed — Safety Risk | 0 | 1
Not completed — Participant unwilling or unable to participate | 0 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nicotinamide | Placebo | Total
Number analyzed (Participants) | 24 | 22 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.56 (8.97) | 72.92 (744) | 73.78 (8.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 14 | 12 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 23 | 21 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 21 | 21 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 22 | 46
Mini-Mental State Examination [Mean (Standard Deviation); unit: units on a scale] — The Mini-Mental State Examination is a brief mental status exam and widely used dementia screening instrument. It evaluates orientation to time and place, memory, attention, language, and visuospatial ability. Range: 0-30; a lower score indicates greater impairment.
  units on a scale | 25.62 (2.87) | 25.5 (3.22) | 25.57 (3.01)

OUTCOME MEASURES:

1. Primary Outcome: Change in P-tau 231
Description: Change in key peptide in cerebrospinal fluid (CSF) from baseline to 48 weeks. Higher phosphorylated tau (p-tau) is associated with a severity of Alzheimer's disease pathology.
Time Frame: Baseline to 48 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Nicotinamide | Placebo
Number analyzed (Participants) | 19 | 19
pg/ml | 4.71 (14.46) | 2.28 (10.55)
Statistical Analysis 1: Comparison: Nicotinamide vs Placebo; Test type: Superiority; p = 0.6096, ANCOVA

2. Primary Outcome: Vital Signs - Weight
Description: Weight in kg was recorded at every study visit (screening, baseline, week 12, week 24, and week 48)
Time Frame: Screening through end of study (week 48)
Population: Numbers analyzed in some rows lower due to missing data (visit not completed, or participant refused measure).
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Nicotinamide | Placebo
Number analyzed (Participants) | 24 | 22
kg
  Screening Visit | 76.39 (12.99) | 68.11 (14.3)
  Baseline Visit | 76.29 (12.57) | 70.05 (11.86)
  Week 12 Visit: number analyzed (Participants) | 22 | 20
  Week 12 Visit | 77.27 (10.86) | 69.36 (12.67)
  Week 24 Visit: number analyzed (Participants) | 20 | 19
  Week 24 Visit | 76.88 (11.49) | 72.22 (11.35)
  Week 48 Visit: number analyzed (Participants) | 21 | 19
  Week 48 Visit | 76.43 (11.96) | 70.27 (12.2)

3. Primary Outcome: Vital Signs - BMI
Description: Body Mass Index (BMI) was recorded at every study visit (screening, baseline, week 12, week 24, and week 48)
Time Frame: Screening through end of study (week 48)
Population: Numbers analyzed in some rows lower due to missing data (visit not completed, or participant refused measure).
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Nicotinamide | Placebo
Number analyzed (Participants) | 24 | 22
kg/m^2
  Screening Visit | 26.35 (4.75) | 24.09 (4.17)
  Baseline Visit | 26.33 (4.69) | 24.85 (3.43)
  Week 12 Visit: number analyzed (Participants) | 22 | 20
  Week 12 Visit | 26.42 (4.51) | 24.72 (3.79)
  Week 24 Visit: number analyzed (Participants) | 20 | 19
  Week 24 Visit | 26.52 (4.56) | 25.08 (3.68)
  Week 48 Visit: number analyzed (Participants) | 21 | 19
  Week 48 Visit | 26.24 (4.75) | 24.68 (3.68)

4. Primary Outcome: Vital Signs - Systolic Blood Pressure
Description: Systolic blood pressure was recorded at every study visit (screening, baseline, week 12, week 24, and week 48)
Time Frame: Screening through end of study (week 48)
Population: Numbers analyzed in some rows lower due to missing data (visit not completed, or participant refused measure).
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nicotinamide | Placebo
Number analyzed (Participants) | 24 | 22
mm Hg
  Screening Visit | 134.67 (19.17) | 126.09 (14.32)
  Baseline Visit | 137.42 (15.99) | 125.41 (17.66)
  Week 12 Visit: number analyzed (Participants) | 22 | 20
  Week 12 Visit | 133.36 (14.91) | 128.05 (18.61)
  Week 24 Visit: number analyzed (Participants) | 20 | 19
  Week 24 Visit | 130.4 (14.04) | 130.16 (13.12)
  Week 48 Visit: number analyzed (Participants) | 21 | 19
  Week 48 Visit | 129.43 (17.76) | 129.37 (17.16)

5. Primary Outcome: Vital Signs - Diastolic Blood Pressure
Description: Diastolic blood pressure was recorded at every study visit (screening, baseline, week 12, week 24, and week 48)
Time Frame: Screening through end of study (week 48)
Population: Numbers analyzed in some rows lower due to missing data (visit not completed, or participant refused measure).
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nicotinamide | Placebo
Number analyzed (Participants) | 24 | 22
mm Hg
  Screening Visit | 75.42 (9.31) | 71.32 (8.97)
  Baseline Visit | 74.21 (11.87) | 70.45 (8.78)
  Week 12 Visit: number analyzed (Participants) | 22 | 20
  Week 12 Visit | 72.45 (7.61) | 71.4 (10.23)
  Week 24 Visit: number analyzed (Participants) | 20 | 19
  Week 24 Visit | 75.2 (7.35) | 71.4 (10.23)
  Week 48 Visit: number analyzed (Participants) | 21 | 19
  Week 48 Visit | 71.9 (10.4) | 69.74 (8.53)

6. Primary Outcome: Vital Signs - Pulse
Description: Pulse rate was recorded at every study visit (screening, baseline, week 12, week 24, and week 48)
Time Frame: Screening through end of study (week 48)
Population: Numbers analyzed in some rows lower due to missing data (visit not completed, or participant refused measure).
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Nicotinamide | Placebo
Number analyzed (Participants) | 24 | 22
bpm
  Screening Visit | 56.42 (6.98) | 62.5 (10.92)
  Baseline Visit | 59.33 (12.85) | 64.91 (8.78)
  Week 12 Visit: number analyzed (Participants) | 22 | 20
  Week 12 Visit | 58.86 (6.14) | 63.45 (11.65)
  Week 24 Visit: number analyzed (Participants) | 20 | 19
  Week 24 Visit | 58.6 (7.42) | 62.26 (8.75)
  Week 48 Visit: number analyzed (Participants) | 21 | 19
  Week 48 Visit | 59.57 (8.33) | 64.84 (12.65)

7. Primary Outcome: Count of Treatment Emergent Adverse Events
Description: Count of treatment emergent adverse events (TEAEs) over the duration of the study period (baseline to 48 weeks).
Time Frame: Baseline to 48 weeks
Measure: Number; unit: events
Arm/Group | Nicotinamide | Placebo
Number analyzed (Participants) | 24 | 22
events | 79 | 71

8. Primary Outcome: Count of Adverse Events by Severity
Description: Count of treatment emergent adverse events (TEAEs) over the duration of the study period (baseline to 48 weeks).
Time Frame: Baseline to 48 weeks
Measure: Number; unit: events
Arm/Group | Nicotinamide | Placebo
Number analyzed (Participants) | 24 | 22
events
  Mild | 49 | 38
  Moderate | 27 | 31
  Severe | 3 | 2
  Total | 79 | 71

9. Primary Outcome: Columbia-Suicide Severity Rating Scale
Description: The Columbia-Suicide Severity Rating Scale (C-SSRS) captures the occurrence, severity, and frequency of suicide-related thoughts and behaviors during the corresponding assessment period. The scale includes suggested questions to elicit the type of information needed to determine if a suicide-related thought or behavior occurred. The number and proportion of subjects with treatment emergent Suicidal ideation or behavior during the study period of (baseline to week 48) will be reported overall and by study arm. Treatment emergent suicidal ideation or behavior is defined as a "yes" answer at any time during treatment to any one of the questions in the ten suicidal ideation and behavior categories (Categories 1- 10) on the C-SSRS. Self-injurious behavior without suicidal intent, while assessed on the C-SSRS, does not form part of this outcome.
Time Frame: Baseline to 48 weeks
Measure: Number; unit: events
Arm/Group | Nicotinamide | Placebo
Number analyzed (Participants) | 24 | 22
events
  Baseline Number of abnormal C-SSRS events | 0 | 3
  Post-baseline number of abnormal C-SSRS events | 1 | 3

10. Primary Outcome: ECG Abnormalities
Description: Count of participants experiencing at least one electrocardiogram (ECG) abnormality.
Time Frame: Baseline to 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotinamide | Placebo
Number analyzed (Participants) | 24 | 22
Participants | 24 | 20

11. Secondary Outcome: Change in ab40
Description: Change in key peptide in cerebrospinal fluid (CSF) from baseline to 48 weeks. Lower ab40 is associated with a greater probability of fibrillar amyloid burden in the brain.
Time Frame: Baseline to 48 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Nicotinamide | Placebo
Number analyzed (Participants) | 19 | 19
pg/ml | 2307 (2516.4) | 1961.1 (4252.97)
Statistical Analysis 1: Comparison: Nicotinamide vs Placebo; Test type: Superiority; p = 0.648, ANCOVA

12. Secondary Outcome: Change in ab42
Description: Change in key peptide in cerebrospinal fluid (CSF) from baseline to 48 weeks. Lower ab42 is associated with a greater probability of fibrillar amyloid burden in the brain.
Time Frame: Baseline to 48 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Nicotinamide | Placebo
Number analyzed (Participants) | 19 | 19
pg/ml | 127.74 (161.54) | 113.79 (321.92)
Statistical Analysis 1: Comparison: Nicotinamide vs Placebo; Test type: Superiority; p = 0.6833, ANCOVA

13. Secondary Outcome: Change in P-tau 181
Description: Change in key peptide in cerebrospinal fluid (CSF) from baseline to 48 weeks. Higher total value is associated with greater severity of Alzheimer's disease pathology.
Time Frame: Baseline to 48 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Nicotinamide | Placebo
Number analyzed (Participants) | 19 | 19
pg/ml | -0.41 (29.83) | -10.43 (41.79)
Statistical Analysis 1: Comparison: Nicotinamide vs Placebo; Test type: Superiority; p = 0.4438, ANCOVA

14. Secondary Outcome: Change in Total Tau
Description: Change in CSF total tau in individuals with mild Alzheimer's disease (AD) dementia or Mild Cognitive Impairment due to AD.
Time Frame: Baseline to 48 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Nicotinamide | Placebo
Number analyzed (Participants) | 19 | 19
pg/ml | -8.42 (228.59) | -60.47 (237.54)
Statistical Analysis 1: Comparison: Nicotinamide vs Placebo; Test type: Superiority; p = 0.7158, ANCOVA

15. Secondary Outcome: Change in Ratio of Total Tau/ab40
Description: Change in ratio of key peptides in cerebrospinal fluid (CSF) from baseline to 48 weeks. A lower ab40/tau ratio is associated with a higher risk of dementia.
Time Frame: Baseline to 48 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Nicotinamide | Placebo
Number analyzed (Participants) | 19 | 19
ratio | -0.02 (0.02) | -0.02 (0.02)
Statistical Analysis 1: Comparison: Nicotinamide vs Placebo; Test type: Superiority; p = 0.93428359, ANCOVA

16. Secondary Outcome: Change in Ratio of Total Tau/ab42
Description: Change in ratio of key peptides in cerebrospinal fluid (CSF) from baseline to 48 weeks. A lower ab42/tau ratio is associated with a higher risk of dementia.
Time Frame: Baseline to 48 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Nicotinamide | Placebo
Number analyzed (Participants) | 19 | 19
ratio | -0.46 (0.56) | -0.5 (0.55)
Statistical Analysis 1: Comparison: Nicotinamide vs Placebo; Test type: Superiority; p = 0.9931, ANCOVA

17. Secondary Outcome: ADASCog-13
Description: ADAS-Cog13 is a structured scale that evaluates memory (immediate and delayed word recall; immediate word recognition), receptive and expressive language, orientation, ideational praxis (preparing a letter for mailing), constructional praxis (copying figures), and attention (number cancellation). Ratings of spoken language, language comprehension, word finding difficulty, and ability to remember test instructions also are obtained. Range: 0-85; higher scores indicate greater impairment.
Time Frame: Baseline to 48 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotinamide | Placebo
Number analyzed (Participants) | 20 | 20
score on a scale | 3.2 (5.72) | 5.16 (7.46)
Statistical Analysis 1: Comparison: Nicotinamide vs Placebo; Test type: Superiority; p = 0.3233, Mixed Models Analysis

18. Secondary Outcome: Activities of Daily Living - Mild Cognitive Impairment
Description: The ADCS-ADL-MCI is a measure of patient functional performance in Alzheimer's Disease and Mild Cognitive Impairment trials. The informant-based questionnaire assesses conduct of basic and instrumental Activities of Daily Living (ADLs). A total of 24 ADLs are evaluated. Scores range from 0 to 53, with higher scores representing more maintained function.
Time Frame: Baseline to 48 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotinamide | Placebo
Number analyzed (Participants) | 20 | 20
score on a scale | -4.05 (4.88) | -1.39 (6.06)
Statistical Analysis 1: Comparison: Nicotinamide vs Placebo; Test type: Superiority; p = 0.1008, Mixed Models Analysis

19. Secondary Outcome: CDR Sum of Boxes
Description: CDR-SB is a composite rating of cognition and everyday function which incorporates both informant input and direct assessment of performance. It assesses through semi-structured interview three cognitive domains (memory, orientation, and judgement/problem solving) and three everyday functional domains (community affairs, home and hobbies, personal care). Level of impairment in each of the six domains is rated from none (score=0) to severe (score=3). The six domain scores are then summed to create the CDR-SB. Range 0-18; higher scores indicate greater impairment.
Time Frame: Baseline to 48 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotinamide | Placebo
Number analyzed (Participants) | 21 | 20
score on a scale | 0.76 (2.03) | 2.18 (2.82)
Statistical Analysis 1: Comparison: Nicotinamide vs Placebo; Test type: Superiority; p = 0.0323, Mixed Models Analysis

20. Primary Outcome: QTC Abnormalities
Description: Count of participants experiencing at least one electrocardiogram (ECG) QT interval abnormality. Abnormal defined as above 460 for men and above 470 for women.
Time Frame: Baseline to 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotinamide | Placebo
Number analyzed (Participants) | 24 | 22
Participants | 2 | 1

21. Primary Outcome: Change in QTC
Description: Average within-subject change in electrocardiogram QT interval.
Time Frame: Baseline to 48 weeks
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Nicotinamide | Placebo
Number analyzed (Participants) | 22 | 21
ms | 6.41 (16.02) | 2.1 (11.85)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from signed consent through the participant duration in the study. The specific time period is from consent through the end of the 48 week double-blind trial. Adverse event information will be collected at every planned and unplanned in-person and telephone visit until 7 (for non-serious AEs) or 30 days (for SAEs) after the last day of study participation.
Arm/Group | Nicotinamide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/22
Serious Adverse Events (participants affected / at risk) | 2/24 | 6/22
Other Adverse Events (participants affected / at risk) | 23/24 | 20/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotinamide (N=24) | Placebo (N=22)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotinamide (N=24) | Placebo (N=22)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (8) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neusea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 0 (0) | 3 (3)
Corona virus infection (Infections and infestations) | 0 (0) | 2 (2)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Gastritis viral (Infections and infestations) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pyuria (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 4 (5) | 4 (5)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 4 (5) | 5 (5)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Antimitochondrial antibody positive (Investigations) | 0 (0) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Blood testosterone decreased (Investigations) | 1 (1) | 0 (0)
Glomerular Ffiltration rate decreased (Investigations) | 1 (1) | 0 (0)
Laboratory test abnormal (Investigations) | 2 (2) | 0 (0)
Urine ketone body present (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Cognitive disorder (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Pleocytosis (Nervous system disorders) | 1 (1) | 0 (0)
Postural tremor (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Syncoper (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Parasomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Penile ulceration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cancer surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Cataract operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Skin neoplasm excision (Surgical and medical procedures) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Labile blood pressure (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2017-12-28): https://cdn.clinicaltrials.gov/large-docs/74/NCT03061474/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT03061474/SAP_001.pdf
  • Informed Consent Form (2021-06-11): https://cdn.clinicaltrials.gov/large-docs/74/NCT03061474/ICF_002.pdf